CLINICAL TRIAL: NCT00435461
Title: A Comparison of Fluticasone Furoate Nasal Spray Versus Oral Fexofenadine in the Treatment of Seasonal Allergic Rhinitis
Brief Title: Fluticasone Furoate Nasal Spray Versus Oral Fexofenadine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: FFU109045
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2017-07

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: once daily; mountain cedar; fexofenadine; allergic rhinitis; fluticasone furoate
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — fluticasone furoate; fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fluticasone furoate and fexofenadine — Fluticasone furoate and fexofenadine

SUMMARY:
The primary objective of this study is to compare the nighttime symptom relief of fluticasone furoate nasal spray and oral fexofenadine

ELIGIBILITY:
Inclusion criteria:

* Informed consent.
* Outpatient.
* Females of child-bearing potential must use appropriate contraception.
* Diagnosis of seasonal allergic rhinitis to mountain cedar.
* Adequate exposure to allergen.
* Able to comply with study procedures.
* Literate.

Exclusion criteria:

* Significant concomitant medical condition.
* Use of corticosteroids, allergy medications, or other medication that affect allergic rhinitis
* Positive pregnancy test.
* Allergy to any component of the investigational product.
* Tobacco use
* Contact lens use
* Has chickenpox or measles or recent exposure
* Other clinical trial drug exposure in last 30 days
* Affiliation with clinic site

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2006-12-20; Primary Completion 2007-02-01 (Actual); Study Completion 2007-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, New Braunfels, Texas
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Andrews C, Martin B, Jacobs R, Toler T, Prillaman B, Philpot E. Efficacy of fluticasone furoate nasal spray versus oral fexofenadine on nighttime sleep disturbance caused by seasonal allergic rhinitis (SAR) nasal symptoms. Ann Allergy Asthma Immunol 2008; 100(1) (Supplement 1):A6 (abstract)
- [Background] Andrews CP, Martin BG, Jacobs RL, Diaz J, Toler WT, Prillaman BA, Dalal AA, Philpot EE. Once-daily fluticasone furoate nasal spray showed greater improvement in nocturnal quality of life in subjects with seasonal allergic rhinitis compared with oral fexofenadine. J Allergy Clin Immunol 2008;121(2) (Supplement 1): S53 (abstract)
- [Background] Andrews CP, Martin BG, Jacobs RL, Mohar DE, Diaz JD, Amar NJ, Kaiser HB, Vandewalker ML, Bernstein J, Toler WT, Prillaman BA, Dalal AA, Lee LA, Philpot EE. Fluticasone furoate nasal spray is more effective than fexofenadine for nighttime symptoms of seasonal allergy. Allergy Asthma Proc. 2009 Mar-Apr;30(2):128-38. doi: 10.2500/aap.2009.30.3204. PMID 19463203
- [Background] Martin BG, Andrews CP, Jacobs R, Mohar D, Toler WT, Prillaman BA, Philpot EE. Once-daily fluticasone furoate nasal spray showed greater improvements in relieving nighttime nasal symptoms and increasing peak nasal inspiratory flow versus oral fexofenadine in subjects with seasonal allergic rhinitis (SAR) J Allergy Clin Immunol 2008;121(2) (Supplement 1): S54-S55 (abstract)
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: FFU109045 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFU109045 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFU109045 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFU109045 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFU109045 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFU109045 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included 5-21 days of screening period followed by two weeks of treatment period and a Follow-up. Participants had to meet five symptom assessment criteria before randomization. Two of these were based on average Nasal Symptom Score assessment and three criteria's were based on the Daytime reflective Nasal Symptom Score (D-rTNSS).
Pre-assignment Details: Total of 1360 participants were planned for enrollment so as to have 951 evaluable participants. A total of 1338 participants were screened and 936 were randomized.
Groups:
- Placebo: Participants received vehicle placebo nasal spray and oral placebo capsule each morning once daily for two weeks following pre-dose symptom assessment.
- FFNS 110 Microgram (mcg): Participants received fluticasone furoate nasal spray (FFNS) 110 mcg and oral placebo capsule each morning once daily for two weeks following pre-dose symptom assessment.
- Fex 180 Milligram (mg): Participants received oral capsule (overencapsulated fexofenadine [Fex] 180 mg oral tablet) and vehicle placebo nasal spray each morning once daily for two weeks following pre-dose symptom assessment.
Period: Overall Study
Arm/Group | Placebo | FFNS 110 Microgram (mcg) | Fex 180 Milligram (mg)
Started | 313 | 312 | 311
Completed | 290 | 298 | 287
Not Completed | 23 | 14 | 24
Not completed — Visit changed to EarlyWithdrawn Visit | 1 | 0 | 0
Not completed — Protocol Violation | 6 | 9 | 10
Not completed — Participant randomized(inadequate score) | 1 | 0 | 0
Not completed — Compliance less than 80 percent | 1 | 0 | 0
Not completed — In error, two study medications switched | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Randomized in error | 1 | 0 | 0
Not completed — Participant could not tolerate symptoms | 0 | 0 | 1
Not completed — Participant could not swallow capsule | 0 | 0 | 1
Not completed — Pregnancy | 2 | 0 | 0
Not completed — Participant moved eDiary,studymedication | 1 | 0 | 0
Not completed — Participant ended study one day early | 1 | 0 | 0
Not completed — Noncompliance with study requirements | 1 | 1 | 1
Not completed — Adverse Event | 1 | 2 | 6
Not completed — Non-Compliance of diary | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- FFNS 110 mcg: Participants received FFNS 110 mcg and oral placebo capsule each morning once daily for two weeks following pre-dose symptom assessment.
- Fex 180 mg: Participants received oral capsule (overencapsulated Fex 180 mg oral tablet) and vehicle placebo nasal spray each morning once daily for two weeks following pre-dose symptom assessment.
- Total: Total of all reporting groups
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg | Total
Number analyzed (Participants) | 313 | 312 | 311 | 936
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (14.39) | 37.8 (13.95) | 39.6 (14.63) | 38.4 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 209 | 199 | 602
  Male | 119 | 103 | 112 | 334
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 22 | 26 | 9 | 57
  American Indian or Alaska Native | 7 | 5 | 6 | 18
  Asian - Central/South Asian Heritage | 3 | 1 | 1 | 5
  Asian - East Asian Heritage | 1 | 2 | 0 | 3
  Asian - Japanese Heritage | 0 | 1 | 0 | 1
  Asian - South East Asian Heritage | 2 | 1 | 2 | 5
  Native Hawaiian or other Pacific Islander | 2 | 1 | 2 | 5
  White/Caucasian/European Heritage | 270 | 268 | 286 | 824
  Mixed Race | 6 | 7 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline Over the Two-week Treatment Period in Nighttime Symptoms Score (NSS)
Description: The NSS is a three-item questionnaire which assesses three aspects of allergic rhinitis symptoms at night which were rated using three 4-point scales, the sum of which comprises NSS. The total score ranged from 0 (best) to 9 (worst). The symptoms were: PM nasal congestion upon awakening (PMNCA) (0- None, 1- Mild, 2- Moderate, 3- Severe), difficulty in going to sleep due to nasal symptoms (DSNS) (0- Not at all, 1- Little, 2- Moderately, 3- Very), and nighttime awakenings due to nasal symptoms (NANS) (0- Not at all, 1- Once, 2- More than once, 3- I felt like I was awake all night). Each participant's Baseline NSS was defined as the average of the NSS calculated for the day of randomization and the three highest NSS scores calculated during the six days immediately prior to the day of randomization. Each participant's average change from Baseline NSS for Weeks 1-2 was the participant's average NSS over the treatment period minus the participant's Baseline NSS.
Time Frame: Baseline (Day 1) and up to 2 Weeks
Population: Intent-to-treat (ITT) population included all participants randomized to double-blind treatment. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 312 | 312 | 309
Scores on a scale
  NSS, Week 1-2 | -1.9 (0.1) | -2.9 (0.1) | -2.0 (0.09)
  PMNCA, Week 1-2 | -0.6 (0.03) | -0.9 (0.03) | -0.6 (0.03)
  NANS, Week 1-2 | -0.7 (0.04) | -1.0 (0.04) | -0.7 (0.03)
  DSNS, Week 1-2 | -0.7 (0.04) | -1.1 (0.04) | -0.8 (0.04)
Statistical Analysis 1: Comparison: FFNS 110 mcg vs Fex 180 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.2 to -0.7], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1, 95% CI 2-sided [-1.2 to -0.7], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Placebo vs Fex 180 mg; Test type: Superiority or Other; p = 0.816, ANCOVA; Mean Difference (Final Values) = -0, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.14

2. Secondary Outcome: Mean Change From Baseline Over the Two-week Treatment Period in Nighttime Reflective Total Nasal Symptom Scores (N-rTNSS) and Component Nasal Symptoms Score
Description: The nighttime reflective assessments were recorded each morning and assessed 4 nasal symptoms (rhinorrhea, nasal congestion, nasal itching, sneezing) at evening and night using a 4-point scale, 0- 'None' (symptom is not present), 1- 'Mild' (sign/symptom present; easily tolerated), 2- 'Moderate' (sign/symptom bothersome but tolerable), 3- 'Severe' (sign/symptom hard to tolerate; interference with activities of daily living). Scores of each of the 4 symptoms were summed for each participant to create a N-rTNSS for each day. The total score ranged from 0 (best) to 12 (worst). Each participant's Baseline total score was average of nighttime total symptom score on day of randomization and 3 highest scores calculated for 6 days immediately prior to day of randomization. Each participant's average change from Baseline nighttime total symptom score for Weeks 1-2 was the participant's average Nighttime total symptom score over the treatment period minus the participant's Baseline score.
Time Frame: Baseline (Day 1) and up to 2 Weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 312 | 312 | 309
Scores on a scale
  TNSS | -2.5 (0.13) | -3.7 (0.14) | -2.7 (0.13)
  Nasal congestion | -0.6 (0.03) | -0.9 (0.04) | -0.7 (0.03)
  Itchy nose | -0.7 (0.04) | -0.9 (0.04) | -0.7 (0.04)
  Runny nose | -0.6 (0.04) | -0.9 (0.04) | -0.7 (0.03)
  Sneezing | -0.7 (0.04) | -1.0 (0.04) | -0.7 (0.04)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-1.6 to -0.9], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: FFNS 110 mcg vs Fex 180 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1, 95% CI 2-sided [-1.4 to -0.7], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Placebo vs Fex 180 mg; Test type: Superiority or Other; p = 0.136, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.18

3. Secondary Outcome: Mean Change From Baseline Over the Two-week Treatment Period in D-rTNSS
Description: The Daytime reflective assessments were recorded each evening and assessed 4 nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing) at evening and night using a 4-point scale, 0- 'None' (symptom is not present), 1- 'Mild' (sign/symptom present; easily tolerated), 2- 'Moderate' (sign/symptom bothersome but tolerable), 3- 'Severe' (sign/symptom hard to tolerate; interference with activities of daily living). The scores of each of the four Daytime symptoms were summed for each participant to create a D-rTNSS for each day. The total score ranged from 0 (best) to 12 (worst). Each participant's Baseline total symptom score was the average of the four highest total symptom score calculated for the seven days immediately prior to the day of randomization. Each participant's average change from Baseline Daytime total symptom score for Weeks 1-2 was the participant's average Daytime total symptom score over the treatment period minus the participants Baseline score.
Time Frame: Baseline (Day 1) and up to 2 Weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 312 | 312 | 309
Scores on a scale
  TNSS | -2.6 (0.13) | -3.7 (0.14) | -3.0 (0.13)
  Nasal congestion | -0.7 (0.04) | -0.9 (0.04) | -0.8 (0.03)
  Itchy nose | -0.7 (0.04) | -1.0 (0.04) | -0.8 (0.04)
  Runny nose | -0.6 (0.04) | -0.9 (0.04) | -0.7 (0.03)
  Sneezing | -0.7 (0.04) | -1.1 (0.04) | -0.9 (0.04)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.5 to -0.7], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: FFNS 110 mcg vs Fex 180 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.2 to -0.4], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Placebo vs Fex 180 mg; Test type: Superiority or Other; p = 0.136, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.19

4. Secondary Outcome: Mean Change From Baseline Over the Two-week Treatment Period in 24-hour Reflective Total Nasal Symptom Scores (24-hour rTNSS) and Component Nasal Score
Description: Daily 24-hour rTNSS was calculated as the average of the corresponding N-rTNSS and D-rTNSS using a 4-point scale where, 0- 'None' (symptom is not present), 1- 'Mild' (sign/symptom present; easily tolerated), 2- 'Moderate' (sign/symptom bothersome but tolerable), 3- 'Severe' (sign/symptom hard to tolerate; interference with activities of daily living). The total score ranged from 0 (best) to 12 (worst). The 24-hour total symptom score for a Day is the average of the daytime total symptom score for that Day and the nighttime score for (D+1). If either component of a given date's 24-hour total symptom score was missing, then the 24-hour total symptom score itself were to be set to missing. Each participant's average change from Baseline 24-hour total symptom score for Weeks 1-2 was the participants average 24-hour total symptom score over the treatment period minus the participant's Baseline score.
Time Frame: Baseline (Day 1) and up to 2 Weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 312 | 312 | 308
Scores on a scale
  TNSS | -2.5 (0.13) | -3.6 (0.14) | -2.8 (0.13)
  Nasal congestion | -0.6 (0.03) | -0.9 (0.04) | -0.7 (0.03)
  Itchy nose | -0.7 (0.04) | -0.9 (0.04) | -0.8 (0.04)
  Runny nose | -0.6 (0.03) | -0.9 (0.04) | -0.7 (0.03)
  Sneezing | -0.7 (0.04) | -1.0 (0.04) | -0.8 (0.04)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.6 to -0.8], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: FFNS 110 mcg vs Fex 180 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.3 to -0.6], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Placebo vs Fex 180 mg; Test type: Superiority or Other; p = 0.136, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.18

5. Secondary Outcome: Mean Change From Baseline Over the Two-week Treatment Period in Nighttime Reflective Total Ocular Symptom Scores (N-rTOSS)
Description: The nighttime reflective assessments were recorded each morning and assessed 3 ocular symptoms (tearing/watering, itching/burning, and redness) at evening and night using a 4-point scale, 0- 'None' (symptom is not present), 1- 'Mild' (sign/symptom present; easily tolerated), 2- 'Moderate' (sign/symptom bothersome but tolerable), 3- 'Severe' (sign/symptom hard to tolerate; interference with activities of daily living). Scores of each of 3 Nighttime symptoms were summed for each participant to create a N-rTOSS for each day. The total score ranged from 0 (best) to 9 (worst). Each participants Baseline total score was average of nighttime total symptom score on day of randomization and the 3 highest scores calculated for 6 days immediately prior to the day of randomization. Each participant's average change from Baseline nighttime total symptom score for Weeks 1-2 was the participant's average Nighttime total symptom score over treatment period minus the participant's Baseline score.
Time Frame: Baseline (Day 1) and up to 2 Weeks
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 312 | 312 | 309
Scores on a scale
  TOSS | -2 (0.11) | -2.5 (0.11) | -2.2 (0.11)
  Eye tearing | -0.7 (0.04) | -0.9 (0.04) | -0.8 (0.04)
  Eye itching | -0.7 (0.04) | -0.9 (0.04) | -0.8 (0.04)
  Eye redness | -0.6 (0.04) | -0.8 (0.04) | -0.7 (0.04)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: FFNS 110 mcg vs Fex 180 mg; Test type: Superiority or Other; p = 0.106, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs Fex 180 mg; Test type: Superiority or Other; p = 0.286, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.15

6. Secondary Outcome: Mean Change From Baseline Over the Two-week Treatment Period in Daytime Reflective Total Ocular Symptom Scores (D-rTOSS)
Description: The Daytime reflective assessments were recorded each evening and assessed the 3 nasal symptoms (tearing/watering, itching/burning, and redness) at evening and night using a 4-point scale where, 0- 'None' (symptom is not present), 1- 'Mild' (sign/symptom present; easily tolerated), 2- 'Moderate' (sign/symptom bothersome but tolerable), 3- 'Severe' (sign/symptom hard to tolerate; interference with activities of daily living). The scores of each of the three Daytime symptoms were summed for each participant to create a D-rTOSS for each day. The total score ranged from 0 (best) to 9 (worst). Each participants Baseline total symptom score was the average of the four highest total symptom score calculated for the seven days immediately prior to the day of randomization. Each participant's average change from Baseline Daytime total symptom score for Weeks 1-2 was the participant's average Daytime total symptom score over the treatment period minus the participant's Baseline score.
Time Frame: Baseline (Day 1) and up to 2 Weeks
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 312 | 312 | 309
Scores on a scale
  TOSS | -2.2 (0.11) | -2.6 (0.11) | -2.4 (0.11)
  Eye tearing | -0.8 (0.04) | -0.9 (0.04) | -0.8 (0.04)
  Eye itching | -0.8 (0.04) | -0.9 (0.04) | -0.9 (0.04)
  Eye redness | -0.7 (0.04) | -0.8 (0.04) | -0.7 (0.04)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Fex 180 mg; Test type: Superiority or Other; p = 0.286, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: FFNS 110 mcg vs Fex 180 mg; Test type: Superiority or Other; p = 0.106, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.15

7. Secondary Outcome: Mean Change From Baseline Over the Two-week Treatment Period in 24-hour Reflective Total Ocular Symptom Scores (24-hour rTOSS)
Description: Daily 24-hour rTOSS was calculated as the average of the corresponding N-rTOSS and D-rTOSS using a 4-point scale, 0- 'None' (symptom is not present), 1- 'Mild' (sign/symptom present; easily tolerated), 2- 'Moderate' (sign/symptom bothersome but tolerable), 3- 'Severe' (sign/symptom hard to tolerate; interference with activities of daily living). The total score ranged from 0 (best) to 9 (worst). The 24-hour total symptom score for a Day is the average of the daytime total symptom score for that Day and the nighttime score for (D+1). If either component of a given date's 24-hour total symptom score was missing, then the 24-hour total symptom score itself was to be set to missing. Each participant's average change from Baseline 24-hour total symptom score for Weeks 1-2 was the participant's average 24-hour total symptom score over the treatment period minus the participant's Baseline score. Baseline is the 4 highest scores calculated for the 7 days prior to Day 1.
Time Frame: Baseline (Day 1) and up to 2 Weeks
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 312 | 312 | 308
Scores on a scale
  TOSS | -2.0 (0.11) | -2.5 (0.11) | -2.2 (0.11)
  Eye tearing | -0.7 (0.04) | -0.9 (0.04) | -0.8 (0.04)
  Eye itching | -0.7 (0.04) | -0.9 (0.04) | -0.8 (0.04)
  Eye redness | -0.7 (0.04) | -0.8 (0.04) | -0.7 (0.04)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Fex 180 mg; Test type: Superiority or Other; p = 0.286, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: FFNS 110 mcg vs Fex 180 mg; Test type: Superiority or Other; p = 0.106, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0], Standard Error of Mean 0.15

8. Secondary Outcome: Mean Change From Baseline Over the Two-week Treatment Period in Pre-dose Instantaneous Total Nasal Symptom Score (Pre-dose iTNSS) and Pre-dose Instantaneous Total Ocular Symptom Scores (Pre-dose iTOSS)
Description: Participants were instructed to score and document their symptoms in an instantaneous manner on a diary card. The instantaneous rating was performed once daily just prior to administering their morning dose. The scores of each of the instantaneous nasal symptoms (nasal congestion, itching, rhinorrhea, and sneezing) and ocular symptoms (tearing/watering, itching/burning, and redness) were summed for each participant to create a iTNSS and iTOSS, respectively using a 4-point scale, 0- 'None' (symptom is not present), 1- 'Mild' (sign/symptom present; easily tolerated), 2- 'Moderate' (sign/symptom bothersome but tolerable), 3- 'Severe' (sign/symptom hard to tolerate; interference with activities of daily living). Total score ranged from 0 (best) to 12 (worst) for iTNSS and 0 (best) to 9 (worst) for iTOSS. Each participant's average change from Baseline iTNSS and iTOSS was participant's average iTNSS and iTOSS total score over the treatment period minus the participant's Baseline score.
Time Frame: Baseline (Day 1) and up to 2 Weeks
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 312 | 312 | 309
Score on a scale
  TNSS | -2.3 (0.13) | -3.6 (0.14) | -2.6 (0.12)
  Pre-dose iTNSS, Nasal congestion | -0.6 (0.03) | -0.8 (0.03) | -0.6 (0.03)
  Pre-dose iTNSS, Itchy nose | -0.7 (0.04) | -1.0 (0.04) | -0.7 (0.04)
  Pre-dose iTNSS, Runny nose | -0.6 (0.04) | -0.9 (0.04) | -0.6 (0.04)
  Pre-dose iTNSS, Sneezing | -0.7 (0.04) | -1.0 (0.04) | -0.7 (0.04)
  TOSS | -1.9 (0.11) | -2.4 (0.12) | -2.2 (0.1)
  Pre-dose iTOSS, Eye tearing | -0.7 (0.04) | -0.9 (0.04) | -0.8 (0.04)
  Pre-dose iTOSS, Eye itching | -0.7 (0.04) | -0.9 (0.04) | -0.8 (0.04)
  Pre-dose iTOSS, Eye redness | -0.6 (0.04) | -0.8 (0.04) | -0.7 (0.04)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg; Pre-dose iTNSS; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-1.7 to -1], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: FFNS 110 mcg vs Fex 180 mg; Pre-dose iTNSS; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.4 to -0.7], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Placebo vs Fex 180 mg; Pre-dose iTNSS; Test type: Superiority or Other; p = 0.193, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.18
Statistical Analysis 4: Comparison: Placebo vs FFNS 110 mcg; Pre-dose iTOSS; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: FFNS 110 mcg vs Fex 180 mg; Pre-dose iTOSS; Test type: Superiority or Other; p = 0.058, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Placebo vs Fex 180 mg; Pre-dose iTOSS; Test type: Superiority or Other; p = 0.16, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to 0], Standard Error of Mean 0.15

9. Secondary Outcome: Mean Change From Baseline Over the Two-week Treatment Period in Peak NasalIinspiratory Flow (PNIF)
Description: PNIF was measured by participants using an In-Check Nasal portable hand-held inspiratory flow meter and face mask. Participants recorded PNIF twice daily (in the morning prior to taking their study medication and in the evening). Three measurements were taken on each occasion and the highest measurement recorded on the electronic diary. Each participant's average change from Baseline PNIF was the participant's average PNIF over the treatment period minus the participant's baseline PNIF.
Time Frame: Baseline (Day 1) and up to 2 Weeks
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Error); unit: Liter(L)/minute (min)
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 313 | 312 | 311
Liter(L)/minute (min)
  Morning PNIF: number analyzed (Participants) | 312 | 312 | 308
  Morning PNIF | 1.7 (0.99) | 9.9 (1.28) | 1.4 (1.18)
  Evening PNIF: number analyzed (Participants) | 312 | 311 | 308
  Evening PNIF | 0.2 (1.12) | 7.1 (1.31) | 1.3 (1.23)
Statistical Analysis 1: Comparison: FFNS 110 mcg vs Fex 180 mg; Morning assessment; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.8, 95% CI 2-sided [5.7 to 11.9], Standard Error of Mean 1.59
Statistical Analysis 2: Comparison: Placebo vs FFNS 110 mcg; Morning assessment; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.4, 95% CI 2-sided [5.3 to 11.5], Standard Error of Mean 1.59
Statistical Analysis 3: Comparison: Placebo vs Fex 180 mg; Morning assessment; Test type: Superiority or Other; p = 0.779, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-3.6 to 2.7], Standard Error of Mean 1.59
Statistical Analysis 4: Comparison: FFNS 110 mcg vs Fex 180 mg; Evening assessment; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [3.1 to 9.6], Standard Error of Mean 1.65
Statistical Analysis 5: Comparison: Placebo vs FFNS 110 mcg; Evening assessment; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7, 95% CI 2-sided [3.8 to 10.3], Standard Error of Mean 1.65
Statistical Analysis 6: Comparison: Placebo vs Fex 180 mg; Evening assessment; Test type: Superiority or Other; p = 0.662, ANCOVA; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-2.5 to 4], Standard Error of Mean 1.65

10. Secondary Outcome: Mean Change From Baseline for Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ)
Description: The NRQLQ is a paper instrument administered on the day of randomization and at Visit 4/Early Withdrawal to assess nocturnal rhinitis-related quality of life. The NRQLQ is a 16-item, self-administered, disease-specific (allergic rhinitis), and quality of life instrument that measures the functional problems most troublesome to patients with nocturnal allergy symptoms over a one-week interval. Each question is scored from 0 to 6 with higher scores indicating more nocturnal impairment. Items are grouped into four domains: Sleep problems, Sleep time problems, Symptoms on waking in the morning and Practical problems. An overall score was calculated from the mean score of all items. Each participant's average change from Baseline NRQLQ score was the participant's average NRQLQ score over the treatment period minus the participant's baseline score.
Time Frame: Baseline (Day 1) and Day 15
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
Number analyzed (Participants) | 313 | 312 | 311
Scores on a scale
  Overall score: number analyzed (Participants) | 308 | 309 | 304
  Overall score | -1.3 (0.08) | -1.9 (0.09) | -1.5 (0.08)
  Sleep problems: number analyzed (Participants) | 308 | 311 | 305
  Sleep problems | -1.2 (0.09) | -1.9 (0.09) | -1.5 (0.09)
  Sleep time problems: number analyzed (Participants) | 308 | 311 | 305
  Sleep time problems | -1.3 (0.09) | -1.9 (0.09) | -1.5 (0.09)
  Symptoms on waking: number analyzed (Participants) | 308 | 309 | 304
  Symptoms on waking | -1.4 (0.09) | -2 (0.1) | -1.5 (0.09)
  Practical problems: number analyzed (Participants) | 308 | 309 | 304
  Practical problems | -1.2 (0.09) | -1.9 (0.1) | -1.6 (0.1)
Statistical Analysis 1: Comparison: FFNS 110 mcg vs Fex 180 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.3], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo vs Fex 180 mg; Test type: Superiority or Other; p = 0.203, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.8 to -0.4], Standard Error of Mean 0.11

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious adverse events (SAEs) were collected from the time the first dose of study medication until the follow up contact (Up to Day 20)
Description: SAEs and non-serious AEs were collected in members of the ITT Population, comprised of all participants randomized to double-blind treatment.
Arm/Group | Placebo | FFNS 110 mcg | Fex 180 mg
All-Cause Mortality (participants affected / at risk) | 0/313 | 0/312 | 0/311
Serious Adverse Events (participants affected / at risk) | 0/313 | 0/312 | 1/311
Other Adverse Events (participants affected / at risk) | 11/313 | 12/312 | 10/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=313) | FFNS 110 mcg (N=312) | Fex 180 mg (N=311)
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=313) | FFNS 110 mcg (N=312) | Fex 180 mg (N=311)
Headache (Nervous system disorders) | 11 | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.